CLINICAL TRIAL: NCT02252003
Title: Development of a New Pain Rating Scale for Children and Validation Against Criteria by Comparison With Faces Pain Scale - Revised (FPS-R) and Visual Analogue Scale (VAS)
Brief Title: Development and Validation of a New Pain Scale for Children
Acronym: NOUNOURS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013.811; 2013-A00849-36 (Registry Identifier: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2014-09-03; First posted 2014-09-29 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Pain
Keywords: Children; Pain; Pain scale evaluation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pain scales testing (Experimental)
  Interventions: Other: Pain scales testing

INTERVENTIONS:
Other: Pain scales testing

SUMMARY:
In clinical practice with young children, gold standard rating scales used to evaluate the pain are VAS (Visual Analogue Scale) and FPS-R (Faces Pain Scale - Revised), which are self-assessment tools. These scales present however certain limitations: the VAS is not applicable if the child does not know how to estimate the distances, as young children, or children with mental retardation. As for FPS-R, it can be frightening for children by the aspect of faces looking like impersonal masks.

For children under 4 years, only hetero-evaluation based on typical behavioral scales as Face Legs Activity Cry Consolability (FLACC) can be used, according to the current recommendations.

We thus wanted to create a new faces scale with teddy bear faces, which are cross-cultural and timeless. Our objective is to validate the new teddy scale in its paper shape on a wide sample of children. We made the hypothesis that the teddy scale would enable to evaluate the pain in the same way that the FPS-R, being better accepted and preferred by children.

The first phase of this study will be to develop the teddy scale with a sample of 30 healthy children from 4 to 11 year-old, having already experienced pain. This stage allows the validation of the images chosen for the scale, to make sure of their relevance and their optimal recognition by the children.

The scale will then be validated with a sample of 218 hospitalized children from 2 to 11 years old, to whom pain is usually evaluated in a systematic way. Children from 4 to 11 years old will have simultaneously the teddy scale, the VAS and the FPS-R. They will be asked to determine which scale they preferred. Children from 2 to 4 years old will have the teddy scale; the FLACC will be filled in by parents.

Tested hypothesis: The discriminating characteristic of the teddy scale is superior to that of the FPS-R scale The validation of the teddy scale will enable to objectify children's pain, to facilitate the decision-making in the choice of the analgesic to prescribe, and to check the efficiency of these decisions. This teddy scale could be used in current practice as a replacement of the FPS-R.

Following this study, we planned to set up a second project in which the teddy scale will be adapted to electronic form (touchpads), to test its adaptability with the children.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated with the French healthcare system
* Agreed to participate in the study, of which parents/ holders of parental authority signed the informed consent form

Scale development phase:

* Children aged from 4 to 11 years at inclusion
* Having already experienced pain

Scale validation phase:

* Children aged from 2 to 11 years old at inclusion
* Hospitalized in one of the Hôpital Femme-Mère-Enfant (HFME) departments
* At risk of presenting pain, that is to whom the pain is usually evaluated in a systematic way

Exclusion Criteria:

* Children among whom the understanding and/or the language is not sufficient to allow a good comprehension of study instructions
* Children participating simultaneously in another interventional research, being able to interfere with the study results

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Pain assessment (4-11 years old) | Baseline
  Children aged 4-11 will be asked to score the pain they feel at that time, using the 3 scales presented in a randomly assigned order. The measure of the correlation between the scores of the 3 pain scales: VAS score (continuing : 0.0 to 10.0), FPS-R score (0,2,4,6,8,10), and teddy scale score (0,2,4,6,8,10) will be evaluated.

SECONDARY OUTCOMES:
Pain assessment (4-11 years old) depending on age. | Baseline
  Children aged 4-11 will be asked to score the pain they feel at that time, using the 3 scales presented in a randomly assigned order. The measure of discriminating characteristics of each scale (teddy scale, FPS-R and VAS), according to the age (continuing age, or in range: 4-6, 6-8 and 8-11) will be performed.
Scale preference (4-11 years old) | Baseline
  The 174 patients (aged 4-11 years old) will be asked to choose the scale they preferred between teddy scale, VAS and FPS-R. The number of times where the teddy scale is preferred will be counted (result expressed in percentage) and compared to the 2 other scales.
Sensibility of change of teddy and FPS-R scales | Baseline
  The sensibility of change (before/after treatment intake) will be measured by the size-effect (mean of the differences divided by the standard deviation before treatment) and by standardized mean responses (mean of the differences divided by the differences standard deviations).
Pain assessment (2-3 years-old) | Baseline
  Children aged 2-3 years old will be asked to score the pain they feel at that time, using the teddy scale while parents will fill up the FLACC scale. The measure of the correlation between scores of the 2 pain scales: teddy scale score (0,2,4,6,8,10) and FLACC score (continuing from 0 to 10), will be performed using statistical models.

CONTACTS AND LOCATIONS:
Overall Officials: Carole VUILLEROT, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de Médecine Physique et Réadaptation Pédiatrique - Hôpital Femme-Mère-Enfant, Bron, France